CLINICAL TRIAL: NCT03385135
Title: Impact of ALLopurInol on Endothelial fuNCtion in diabEtic Patients Affected With Coronary Artery Disease
Brief Title: Allopurinol and Endothelial Function in Diabetic CAD Patients
Acronym: ALLIENCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Kasbaoui sami, Principal Investigator, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALLIENCE
Record Dates: First submitted 2017-12-14; First posted 2017-12-28 (Actual); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Diabetes Mellitus; Coronary Artery Disease
Keywords: allopurinol; coronary artery disease; diabetes; endothelial function
MeSH Terms: conditions — Diabetes Mellitus; Coronary Artery Disease | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Allopurinol group (Active Comparator): Optimal medical therapy associated with allopurinol. The dose of allopurinol is 300 mg for 4 weeks then 600 mg for 4 weeks
  Interventions: Drug: Allopurinol
- No Allopurinol group (No Intervention): Optimal medical therapy alone

INTERVENTIONS:
Drug: Allopurinol — 300 mg for 4 weeks then 600 mg for 4 weeks in the active group
  Other Names: Optimal Medical Therapy
  Arms: Allopurinol group

SUMMARY:
This is a randomized trial assessing the impact of allopurinol on endothelial function in optimally treated diabetic patients with coronary artery disease. After initial screening, subjects were randomized to receive either optimal medical therapy (OMT) + allopurinol or OMT alone for 8 weeks. The dose of allopurinol was 300 mg for 4 weeks and 600 mg for 4 weeks with a 4-weekly check on hematology and biochemistry

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type 2
* Known coronary artery disease with previous percutaneous coronary intervention and optimal medical therapy for at least one month

Exclusion Criteria:

* Pregnant or breast- feeding women
* creatinine clearance <60ml/min
* Known history of gout disease or ongoing treatment with allopurinol
* Allergy to allopurinol
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Endothelium-dependent vasodilation | 2 months
  Brachial Artery Flow-Mediated dilation (FMD)

SECONDARY OUTCOMES:
Endothelium-independent vasodilation | 2 months
  Changes in brachial artery diameter in response to nitrates
Quality of Life (QoL) | 2 months
  Seattle Angina Questionnaire: a scale that quantifies patients' physical limitations caused by angina, the frequency of and recent changes in their symptoms, their satisfaction with treatment, and the degree to which they perceive their disease to affect their quality of life. Each scale is transformed to a score of 0 to 100, where higher scores indicate better function (eg, less physical limitation, less angina, and better quality of life).
Major adverse cardiac events (MACE) | 2 months
  composite of cardiac death, non fatal myocardial infarction and unplanned coronary revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Salem Kachboura, MD, Study Chair — Cardiology Department, Abderrahmen Mami Hospital, 2008, Ariana
Locations (1):
- Cardiology Department, Abderrahmen Mami Hospital, Aryanah, Tunisia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol